CLINICAL TRIAL: NCT07188467
Title: Implementing a Scalable Mental Health Intervention for International Students: A Pilot Study of Digitized Self-Help Plus
Brief Title: Testing Adapted Self-Help Plus (SH+) for Stress and Well-Being in International Students at a U.S. University
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The New School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SH2025-001
Record Dates: First submitted 2025-09-16; First posted 2025-09-23 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Stress, Psychological; Depression and/or Anxiety in the Mild-to-moderate Range; Loneliness; Adjustment, Psychological
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Self-Help Plus (SH+) Workshop (Experimental): Participants will attend a two-day in-person workshop featuring digitized SH+ materials. The workshop includes animated videos, guided stress management exercises, and group discussions.
  Interventions: Behavioral: Digitized SH+

INTERVENTIONS:
Behavioral: Digitized SH+ — Digitized SH+ is a group-based, stress management program (adapted from the original Self-Help Plus intervention developed by the World Health Organization), that utilizes animated videos and group discussions to teach participants skills such as Grounding, Unhooking (from difficult thoughts), Being Kind (to self and others), Identifying Values, and Making Room for Difficult Thoughts and Feelings.

SUMMARY:
The goal of this clinical trial is to learn if an adapted version of Self-Help Plus (SH+), a stress management program developed by the World Health Organization, can reduce stress and improve well-being in international students at a U.S. university. The main questions it aims to answer are:

Does SH+ reduce perceived stress, anxiety, and depressive symptoms in international students? Does SH+ improve feelings of social support, self-efficacy, and adjustment in a new cultural environment?

Participants will:

Attend a two-day in-person workshop that includes animated videos, interactive activities, and group discussions.

Complete three surveys (before the workshop, right after, and six weeks later) about stress, mood, and well-being.

Optionally, take part in a short interview to share feedback about their experience.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled as an international student at The New School
* Age 18 years or older
* Willing to provide informed consent and complete study assessments
* Score of ≥3 on the PHQ-4, indicating at least mild distress
* Sufficient English proficiency to comprehend intervention materials

Exclusion Criteria:

* Severe psychiatric conditions requiring immediate intervention (e.g., active psychosis, severe mood disorders)
* Visual, hearing, or neurocognitive impairments that prevent engagement with the intervention
* Having an advanced degree in psychology or mental health-related fields (to prevent prior knowledge bias)
* Score of 2 or higher on PHQ-4 Item 3 or Item 4 (frequent thoughts of self-harm or severe distress)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-07 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress Scale (PSS-10) | Change from baseline to 6-week follow-up
  Self-reported perceived stress levels. Higher scores indicate greater perceived stress.
  Range: 0-40 Higher scores= worse outcome (greater perceived stress) Cutoffs: 0-13 low, 14-26 moderate, 27-40 high
Patient Health Questionnaire (PHQ-9) | Change from baseline to 6-week follow-up
  Range: 0-27 Higher scores = worse outcome (greater depression severity). Cutoffs: 1-4 minimal, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe.
General Anxiety Disorder (GAD-7) | Change from baseline to 6-week follow-up
  Range: 0-21 Higher scores = worse outcome (greater anxiety severity) Cutoffs: 0-4 minimal, 5-9 mild, 10-14 moderate, 15-21 severe

SECONDARY OUTCOMES:
Self-Measure for Loneliness (UCLA Loneliness Scale) | Change from baseline to 6-week follow-up
  Range: 0-60 (20 items, scored 0-3) Higher scores = worse outcome (greater loneliness/social isolation).
Social Support (SSQ) | Change from baseline to 6-week follow-up
  Range varies (depends on individual): self-reported number of people available for support + satisfaction rating).
  Higher scores = better outcome (greater perceived support and satisfaction).
Self-Efficacy (General Self-Efficacy Scale) | Change from baseline to 6-week follow-up
  Range: 10-40 (10 items, scored 1-4). Higher scores = better outcome (greater self-efficacy/confidence in coping).
Psychological Adjustment (BASE-6) | Change from baseline to 6-week follow-up
  Range: 6-42 (six items, each scored 1-7). Higher scores = worse outcome (greater emotional distress and adjustment difficulty).

CONTACTS AND LOCATIONS:
Overall Officials: Adam D Brown, PhD, Principal Investigator — The New School, Center for Global Mental Health
Locations (1):
- The New School, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No